CLINICAL TRIAL: NCT00144924
Title: Recovery After Open Versus Laparoscopic Pyloromyotomy for Pyloric Stenosis: a Double-blind Multicentre Randomised Controlled Trial
Brief Title: Open vs Laparoscopic Pyloromyotomy for Pyloric Stenosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The aim was to recruit 200 infants (100 per group); however, the data monitoring and ethics committee recommended halting the trial before full recruitment because of significant treatment benefit in one group at interim analysis.
Sponsor: Institute of Child Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 03SG45
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Pyloric Stenosis
MeSH Terms: conditions — Pyloric Stenosis

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- laparoscopic pyloromyotomy (Experimental)
  Interventions: Procedure: laparoscopy pyloromyotomy
- open pyloromyotomy (Active Comparator)
  Interventions: Procedure: open pyloromytomy

INTERVENTIONS:
Procedure: laparoscopy pyloromyotomy — laparoscopic pyloromyotomy
  Arms: laparoscopic pyloromyotomy
Procedure: open pyloromytomy — open pyloromyotomy
  Arms: open pyloromyotomy

SUMMARY:
Comparison of open and laparoscopic pyloromyotomy

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of infantile hypertrophic pyloric stenosis

Exclusion Criteria:

* Presence of co-existing congenital or chromosomal abnormality
* The need to perform any additional procedure at the time of pylotomyotomy
* Failure to receive informed consent

Ages: 0 Months to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2004-06 (Actual); Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Time to full feeds | 6 weeks
Post operative length of stay | 6 weeks
Episodes of post-operative vomiting | 24h

SECONDARY OUTCOMES:
Peri-operative complications | 24h
Post-operative complications | 6 weeks
Anaesthetic time | 24h
Operating time | 24h
Post-operative pain and analgesia requirements | 6 weeks
Cosmetic outcome | 6 weeks
Total in-hospital costs | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Hall, Mr, Principal Investigator — Institute of Child Health
Locations (1):
- Institute of Child Health/Great Ormond Street Hospital, London, United Kingdom

REFERENCES:
- [Result] Hall NJ, Pacilli M, Eaton S, Reblock K, Gaines BA, Pastor A, Langer JC, Koivusalo AI, Pakarinen MP, Stroedter L, Beyerlein S, Haddad M, Clarke S, Ford H, Pierro A. Recovery after open versus laparoscopic pyloromyotomy for pyloric stenosis: a double-blind multicentre randomised controlled trial. Lancet. 2009 Jan 31;373(9661):390-8. doi: 10.1016/S0140-6736(09)60006-4. Epub 2009 Jan 18. PMID 19155060
- [Derived] Carrington EV, Hall NJ, Pacilli M, Drake DP, Curry JI, Kiely EM, De Coppi P, Pierro A, Eaton S. Cost-effectiveness of laparoscopic versus open pyloromyotomy. J Surg Res. 2012 Nov;178(1):315-20. doi: 10.1016/j.jss.2012.01.031. Epub 2012 Mar 27. PMID 22480835